CLINICAL TRIAL: NCT04139018
Title: Efficacy of a Timolol Gel in the Care for Epistaxis in Patients With Hereditary Hemorrhagic Telangiectasia: A Double-Blinded, Randomized Controlled Trial
Brief Title: Timolol Gel for Epistaxis in Hereditary Hemorrhagic Telangiectasia
Acronym: ETIC-HHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Professor and Vice Chair for Research, Department of Otolaryngology - Head and Neck Surgery, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201908160
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Results first posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-07

CONDITIONS: Hereditary Hemorrhagic Telangiectasia
Keywords: Epistaxis
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Timolol Gel Arm (Experimental): Participants in the timolol gel arm (active medication arm) will receive timolol nasal gel 0.1% with 0.5 mL applied to each nostril twice daily via a syringe that will amount to a 2 mg total daily dose.
  Interventions: Drug: Timolol Gel
- Placebo Gel Arm (Placebo Comparator): Participants in the placebo gel arm will receive the gel itself with no active medication.
  Interventions: Drug: Placebo Gel

INTERVENTIONS:
Drug: Timolol Gel — Timolol nasal gel 0.1% will be prepared with a poloxamer gel (combination of poloxamer 188 and 407; pH adjusted to 4.5-6.5) and 0.5 ml applied to each nostril twice daily. The total daily dose would amount to 2 mg.
  Arms: Timolol Gel Arm
Drug: Placebo Gel — Placebo gel is prepared with poloxamers and no active ingredients.
  Arms: Placebo Gel Arm

SUMMARY:
This study is a double-blinded, randomized controlled trial to evaluate the efficacy of an intranasal topical timolol gel in the care for epistaxis in adults with hereditary hemorrhagic telangiectasia.

DETAILED DESCRIPTION:
This study is a double-blinded, placebo-controlled, 8-week randomized clinical trial investigating the efficacy of timolol gel in the management of epistaxis in adults with HHT.

The Specific Aims are to determine in adults with HHT-associated epistaxis:

1. If topical timolol gel is more effective than placebo in reducing the frequency and severity of epistaxis.
2. If topical timolol gel is more effective than placebo in improving hemoglobin levels.
3. The frequency of adverse events, side effects, and safety profile of topical timolol gel delivered to the nasal mucosa.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 20 and older
2. Confirmed clinical (meeting at least 3 of the 4 Curaçao Criteria) or genetic diagnosis of HHT
3. Epistaxis Severity Score (ESS) ≥ 4 and 2 or more nosebleeds per week with a cumulative nosebleed duration of at least 5 minutes per week
4. Stable nasal hygiene and medical regimen for preceding 1 month
5. Stable epistaxis pattern over the preceding 3 months

Exclusion Criteria:

1. Contraindications for systemic β adrenergic blocker administration

   1. Hypersensitivity to β adrenergic blockers
   2. Asthma or bronchospasm
   3. Congestive heart failure with LVEF <40%
   4. Hereditary pulmonary arterial hypertension
   5. Baseline bradycardia (HR <55 beats per minute)
   6. Sick Sinus Syndrome
   7. 2nd or 3rd degree heart block, left or right bundle branch block, or bifasicular block
   8. Uncontrolled diabetes mellitus (most recent HbA1c >9%) or diabetic ketoacidosis within last 6 months
   9. Hypotension (systolic blood pressure < 90)
2. Known hypersensitivity to timolol
3. Severe peripheral circulatory disturbances (Raynaud phenomenon)
4. Known intermediate or poor metabolizer variant of the liver enzyme CYP2D6
5. Current use of any of the following known strong CYP2D6 inhibitors: fluoxetine (Prozac), paroxetine (Paxil), bupropion (Welbutrin), quinidine, quinine, ritonavir (Norvir), and terbinafine (Lamisil)
6. Current use of the following other drugs known to pharmacodynamically interact with timolol: diltiazem, verapamil, digoxin, digitalis, propafenone, disopyramide, clonidine, flecainide, or lidocaine
7. Patients currently treated or who plan to initiate treatment with β-blockers
8. Use of any anti-angiogenic medication in the last month prior to recruitment, including bevacizumab, pazopanib, thalidomide, or lenalidomide
9. Illicit drug use, except marijuana
10. Known pheochromocytoma
11. Use of anticoagulants, antiplatelet, or fibrinolytic therapies within the last month prior to recruitment, except for low-dose (81 mg or less) of aspirin
12. Pregnancy or planned pregnancy in the next 6 months or currently breastfeeding
13. Inability to read or understand English
14. Inability to complete 8 weeks of therapy for any reason

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Derived] Peterson AM, Lee JJ, Kallogjeri D, Schneider JS, Chakinala MM, Piccirillo JF. Efficacy of Timolol in a Novel Intranasal Thermosensitive Gel for Hereditary Hemorrhagic Telangiectasia-Associated Epistaxis: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2020 Nov 1;146(11):1006-1014. doi: 10.1001/jamaoto.2020.3025. PMID 32940653

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from October 2019 through March 2020 at Washington University HHT Center of Excellence
Pre-assignment Details: 272 participants total were assessed for eligibility; 245 met exclusion criteria
Period: Overall Study
Arm/Group | Timolol Gel Arm | Placebo Gel Arm
Started | 14 | 13
Completed | 11 | 12
Not Completed | 3 | 1
Not completed — Screen fail | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Timolol Gel Arm | Placebo Gel Arm | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Median (Full Range); unit: years] | 58 [20 to 76] | 52 [30 to 65] | 55 [20 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 4 | 9 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 14 | 11 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27
Hypertension [Count of Participants; unit: Participants] | 4 | 2 | 6
Seasonal Allergies [Count of Participants; unit: Participants] | 9 | 9 | 18
Comorbidity Status [Count of Participants; unit: Participants]
  None | 9 | 8 | 17
  Mild | 3 | 4 | 7
  Moderate | 1 | 0 | 1
  Severe | 1 | 1 | 2
Baseline Clinical Global Impression - Severity [Count of Participants; unit: Participants] — Measures severity of epistaxis on a 5-point Likert scale from "No problem" to "Problem as bad as it could be"
  Participants
    No Problem | 0 | 0 | 0
    Mild Problem | 3 | 4 | 7
    Moderate/Severe Problem | 10 | 5 | 15
    Problem as bad as it could be | 0 | 0 | 0
    Unknown | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Assisted Epistaxis Severity Scale (aESS) Score From Baseline at 8 Week Follow-up
Description: Assessment of epistaxis severity will be obtained by the validated instrument, the Epistaxis Severity Score (ESS). To complete the ESS, patients are asked to consider typical symptoms over the previous 3 months. The ESS contains 6 items - frequency, duration, and intensity of nosebleeds, whether patient has sought medication attention, whether patient is anemic, and whether patient has received a blood transfusion. The overall score ranges from 0 to 10, with severity of nosebleed based on score graded as None composite score of 0-1, Mild 1-4, Moderate 4-7, and Severe as 7-10.The minimal important difference noticeable by both patients and clinicians in the ESS scoring system is estimated as a change of 0.71. The scoring and MCID of the aESS is the same as the ESS.
  The aESS references a participant's epistaxis over the past 1 month, and the change in aESS was calculated as the aESS score at 8 weeks minus the aESS score at baseline.
Time Frame: Baseline to 8-week follow-up
Population: Analysis was used with intention-to-treat principles, so all patients enrolled with baseline data were included. Note: the screen fail participant within the timolol gel arm had no baseline data say they were excluded from the analysis.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Timolol Gel Arm | Placebo Gel Arm
Number analyzed (Participants) | 13 | 13
units on a scale | 2.32 [0.22 to 5.97] | 1.96 [-0.91 to 5.98]

2. Secondary Outcome: Number of Participants With Improved Response on Clinical Global Impression - Improvement (CGI-I) Scale
Description: CGI-I is a global rating of improvement scale, which requires subjects to rate their degree of improvement on a seven-point scale: "Compared to your condition at admission to the project [prior to medication initiation], how would you rate your overall response: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment."
Time Frame: Scores at 8-week follow-up only
Measure: Count of Participants; unit: Participants
Arm/Group | Timolol Gel Arm | Placebo Gel Arm
Number analyzed (Participants) | 11 | 12
Participants
  No Change | 0 | 1
  Slightly Improved | 4 | 3
  Much Improved | 7 | 8

ADVERSE EVENTS:
Time Frame: Adverse events collected throughout the whole duration of the study and assessed multiple times throughout a participant's 8 weeks of intervention.
Arm/Group | Timolol Gel Arm | Placebo Gel Arm
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 7/14 | 3/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Timolol Gel Arm (N=14) | Placebo Gel Arm (N=13)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dizziness (Vascular disorders) | 1 | 0
Nasal congestion (General disorders) | 3 | 0
Headache (General disorders) | 1 | 1
Rhinorrhea (General disorders) | 1 | 0
Nausea (General disorders) | 1 | 0
Bad taste of medication (General disorders) | 1 | 0
Sore throat (General disorders) | 0 | 1
Irritation upon applying gel (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT04139018/Prot_SAP_001.pdf